CLINICAL TRIAL: NCT04912635
Title: Evaluation of a Health Dashboard Intervention to Improve Engagement With CPAP Therapy in PAP-Naïve Patients: Project Neo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ResMed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: DHT-20-06-01
Record Dates: First submitted 2021-05-28; First posted 2021-06-03 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-05

CONDITIONS: Sleep Apnea, Obstructive
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention)
- Intervention (Experimental)
  Interventions: Other: Neo App

INTERVENTIONS:
Other: Neo App — Neo is a smartphone-based dashboard application that utilizes concepts from behavioral science and health psychology to support patients to improve their adherence to therapy. This is done through behavior change techniques and intervention functions (Michie, Atkins & West, 2014). This app is designed to prompt participants' self-regulation of lifestyle and health behaviors, to support adherence to therapy. Such self-regulation of lifestyle behaviors is informed by presenting health metric data (through wearables, myAir (biofeedback) and self-report), in an easy to understand dashboard platform on the app. Participants will be asked to use their PAP device (as normal), use a Withings blood pressure cuff and activity monitor. This data is brought into the Neo app through an API Exchange gateway. This data will be presented to the participant and communicated in an easy to understand way.
  Arms: Intervention

SUMMARY:
This is a prospective, open-label study to evaluate the effectiveness of providing a dashboard with merged health metrics of CPAP (continuous positive airway pressure/ PAP) usage, self-reported sleepiness, blood pressure (BP) and activity (steps).

ELIGIBILITY:
Inclusion Criteria:

* Participant is at least 18 years old.
* Participant is using a ResMed AirSense 10 device and ResMed myAir mobile app.
* Participant has been using CPAP therapy for less than 2 weeks.
* Participant has been enrolled in myAir for less than 2 weeks.
* Participants have self-reported resistant hypertension and they take 3 or more drugs to treat their hypertension.
* Participant owns a mobile device compatible with the Neo app (Android Jelly Bean, v16, 4.1.x or newer, and iOS 8 or newer)
* Participant is somewhat to fairly confident about being able to use Bluetooth connected devices and apps
* Participant consents to download the Neo app, Withings app, create a Withings account, and sync Withings data to ResMed's Project Neo.
* Willing and able to give informed consent
* Can read and comprehend written and spoken English

Exclusion Criteria:

* Are participating in another app-based research study
* Cannot participate for the full duration of the study (at least 45 days)
* Unable to read or write English
* Participant is pregnant
* Participant is on Medicare

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2020-09-25 (Actual); Primary Completion 2020-12-19 (Actual); Study Completion 2021-03-25 (Actual)

PRIMARY OUTCOMES:
Mean CPAP use hours | 6 weeks
  Mean PAP use hours (mean hours per day) at 6 weeks following enrollment into the study compared to the control group.

SECONDARY OUTCOMES:
App Use | 6 weeks
  Percentage of participants that actively use the Neo app as determined by daily active users, weekly active users and time spent in the app.

CONTACTS AND LOCATIONS:
Locations (1):
- ResMed, Bella Vista, New South Wales, Australia